CLINICAL TRIAL: NCT02285829
Title: Determination of TOF Test Threshold for Obtaining Reliable Pedicle Screw Stimulation Test During Lumbar Spine Surgery
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01568
Record Dates: First submitted 2014-10-27; First posted 2014-11-07 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Rocuronium; cisatracurium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- T4/T1=0.1-0.25: Continuous infusion will commence at the lower dose indicated (0.01mg/kg/min IV for Rocuronium, 0.5 µg/kg/min for Cisatracurium ), and TOF ratios will be monitored every 20 seconds. T4/T1 ratio of quantitative TOF test will be measured, prior pedicle screw stimulation test. When TOF ratio ranges 0.1-0.25, values of pedicle screw stimulation test will be then measured and recorded in milliamps (mA) after TOF test is performed.
  Interventions: Drug: Rocuronium Bromide, Cisatracurium Besylate
- T4/T1=0.25-0.50: Continuous infusion will commence at the lower dose indicated (0.01mg/kg/min IV for Rocuronium Bromide, 0.5 µg/kg/min for Cisatracurium Besylate ), and TOF ratios will be monitored every 20 seconds. T4/T1 ratio of quantitative TOF test will be measured, prior pedicle screw stimulation test. When TOF ratio ranges 0.25-0.50, values of pedicle screw stimulation test will be then measured and recorded in milliamps (mA) after TOF test is performed.
  Interventions: Drug: Rocuronium Bromide, Cisatracurium Besylate
- T4/T1=0.50-0.75: Continuous infusion will commence at the lower dose indicated (0.01mg/kg/min IV for Rocuronium Bromide, 0.5 µg/kg/min for Cisatracurium Besylate ), and TOF ratios will be monitored every 20 seconds. T4/T1 ratio of quantitative TOF test will be measured, prior pedicle screw stimulation test. When TOF ratio ranges 0.50-0.75, values of pedicle screw stimulation test will be then measured and recorded in milliamps (mA) after TOF test is performed.
  Interventions: Drug: Rocuronium Bromide, Cisatracurium Besylate
- T4/T1=0.75-0.90: Continuous infusion will commence at the lower dose indicated (0.01mg/kg/min IV for Rocuronium Bromide, 0.5 µg/kg/min for Cisatracurium Besylate ), and TOF ratios will be monitored every 20 seconds. T4/T1 ratio of quantitative TOF test will be measured, prior pedicle screw stimulation test. When TOF ratio ranges 0.75-0.90, values of pedicle screw stimulation test will be then measured and recorded in milliamps (mA) after TOF test is performed.
  Interventions: Drug: Rocuronium Bromide, Cisatracurium Besylate

INTERVENTIONS:
Drug: Rocuronium Bromide, Cisatracurium Besylate — Both Rocuronium Bromide and Cisatracurium Besylate are administered intravenously following induction of anesthesia initially by bolus, and subsequently re-bolused or administered in continuous infusion as clinically indicated to maintain muscle relaxation. Initial doses of Rocuronium range from 0.45 to 1.2 mg/kg IV, and doses for continuous infusion range from 0.01-0.012 mg/kg/min IV. Initial doses of Cisatracurium range from 0.15 to 0.2 mg/kg, and doses for continuous infusion range from 0.5 to 3 µg/kg/min. Following recovery and baseline screw stimulation at TOF >0.9, the dosing regimen for this study will rely on restarting a continuous infusion, and adjusting the infusion until the desired TOF ratios are reached. Following screw stimulations and data collection, the infusion will be terminated, and neuromuscular blockade allowed to recover.
  Other Names: Zemurone, Nimbex

SUMMARY:
During lumbar spine fusion surgery intraoperative neurophysiological monitoring is in routine use for prevention of possible nerve injuries during placement of screw into pedicle. Pedicle screw stimulation test is performed to assess if screw placement is encroaching on the nerve roots. Relative distance between the pedicle screw and the neighbouring root can be estimated by the intensity of the current required to activate the root and appropriate muscle. A properly placed screw can be distinguished from those perforating the pedicle wall by its higher minimum level of electrical current needed to elicit a muscle response. The minimum level is deemed as threshold. This test is based on compound muscle action potential (CMAP) and use of neuromuscular blocking agents (NMBA) should be avoided because of possible cause of false negative results of screw stimulation test. Neuromuscular blocking agents, which are in routine use during anesthesia, will have effect on muscle action potential. When NMBA are used current stimulus will depolarize the same number of axons and the associated muscle response will be present but of lower amplitude because some percentage of motor fibers will be blocked by activity of NMBA. At this point, stronger stimulus is needed to recruit additional axons/muscle fibers , and hence, the measured threshold is elevated.

Train of four (TOF) test is method used to determine level of neuromuscular blockade, by stimulation of peripheral nerve and following induced muscle contractions. Interpretation of muscle contractions may be by subjective (visual) or objective (quantitative) method. Quantitative TOF test may be used prior screw stimulation test by calculating T4/T1 ratio and obtaining quantitative value which shows level of neuromuscular blockade. Residual neuromuscular blockade may be present before screw stimulation test, and effect on accuracy of this test in this situation was not clearly investigated in recent studies.

The purpose of this study would be to determine changes of screw stimulation thresholds under different range of neuromuscular blockade.Therefore, acceptable neuromuscular blockade threshold (determined by TOF test) acceptable for obtaining reliable screw stimulation test should be determined. Screw stimulation test may be performed when neuromuscular blockade is absent and compared to repeated screw stimulation test when neuromuscular blockade is present. Different levels of neuromuscular blockade may provide different results on screw stimulation test, so if difference is statistically significant, induced neuromuscular blockade level may be set as threshold value, acceptable for obtaining reliable testing results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing lumbar spine fusion surgery with neurophysiologic intraoperative monitoring when pedicle screw stimulation test is performed.
* Subjects of both gender
* Age 18-85
* With diagnosis of lumbar spinal stenosis.
* All subjects capable of giving informed consent in order to be included for the study.

Exclusion Criteria:

* Subjects with medical history of presence of neuromuscular disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing elective lumbar spine fusion surgery
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Train of four (TOF) test | TOF test measure will be performed during the day of surgery prior pedicle screw stimulation test
  T4/T1 ratio will be determined and measured prior pedicle screw stimulation test, during lumbar spine surgery. Data will be obtained and followed from participants during one day, while surgery is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Beric, MD, Principal Investigator — Neurologist
Locations (1):
- NYU Langone Medical Center, Hospital for Joint Diseases, New York, New York, United States